CLINICAL TRIAL: NCT04302857
Title: Pilot Study for Establishing Perioperative Tractography at Leipzig University Neurosurgery
Brief Title: Tractography Pilot Study Leipzig
Status: Completed | Type: Observational
Sponsor: Tim Wende (Other)
Responsible Party: Sponsor-Investigator, Tim Wende, MD, University of Leipzig
Organization: University of Leipzig (Other)
Other Study IDs: 322/19-ek
Record Dates: First submitted 2020-03-06; First posted 2020-03-10 (Actual); Last update posted 2022-06-10 (Actual); Status verified 2022-06

CONDITIONS: Intracranial Neoplasm
MeSH Terms: conditions — Brain Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: routine MRI — MRI with routine DTI sequence

SUMMARY:
In this pilot study participants will undergo routine magnetic resonance imaging and routine neurosurgical care. By prospectively collecting data from both MRI and patient records we want to investigate biomarkers derived from tractography and diffusion tensor imaging to predict rehabilitation potential.

DETAILED DESCRIPTION:
Patients will undergo MRI before and after surgery with DTI. With CSD-tractography, fiber bundles and their volumes will be identified. By measuring fractional anisotropy (FA) within these volumes, a correlation with clinical outcome and recovery will be tested. Also, FA frequency distributions will be used to describe white matter integrity and to thereby improve future tractography algorithms. Fiber bundles of interest will be the arcuate fascicle (AF), the corticospinal tract (CST), frontal aslant tract (FAT), the inferior fronto-occipital fascicle (IFOF), the inferior longitudinal fascicle (ILF) and the uncinate fascicle (UF).

ELIGIBILITY:
Inclusion Criteria:

* intracranial lesion
* elective neurosurgical procedure

Exclusion Criteria:

* MRI not applicable
* cerebral ischemia during study period
* pregnancy during study period
* encephalitis during study period
* spontaneous intracerebral hemorrhage during study period

Ages: 18 Years to 75 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Standard cohort of neurosurgical patients
Sampling Method: Non-Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2020-01-01 (Actual); Primary Completion 2021-12-31 (Actual); Study Completion 2021-12-31 (Actual)

PRIMARY OUTCOMES:
Neurological Performance | three months
  Neurological Performance Score (NPS)

CONTACTS AND LOCATIONS:
Overall Officials: Jürgen Meixensberger, MD, Study Chair — University of Leipzig
Locations (1):
- Leipzig University Hospital, Department of Neurosurgery, Leipzig, Saxony, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Wende T, Hoffmann A, Scherlach C, Kasper J, Sander C, Arlt F, Dietel E, Stockert A, Meixensberger J, Prasse G. Preserved White Matter Integrity and Recovery After Brain Tumor Surgery: A Prospective Pilot Study on the Frontal Aslant Tract. Brain Connect. 2023 Dec;13(10):589-597. doi: 10.1089/brain.2023.0033. Epub 2023 Oct 19. PMID 37646398